CLINICAL TRIAL: NCT01820858
Title: A Multicenter, Prospective, Randomized Trial of the Efficacy and Safety of the Postoperative Adjuvant Treatment in Patients With High-risk Stage I Endometrial Carcinoma
Brief Title: The Efficacy and Safety of the Postoperative Adjuvant Treatment in Patients With High-risk Stage I Endometrial Carcinoma
Acronym: EC-01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ding Ma (Other)
Collaborators: Shandong University (Other); Huazhong University of Science and Technology (Other); Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Ding Ma, Director of the department of Obstetrics and Gynecology, Tongji Hospital, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-GYN/EC-01
Record Dates: First submitted 2013-03-20; First posted 2013-03-29 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant Chemotherapy (Experimental): Paclitaxel: 175 mg/m(2) intravenously (IV); followed by Paraplatin (Carboplatin Injection) AUC=5 IV. 3-6 cycles as necessary.
  Interventions: Drug: Paclitaxel; Drug: Paraplatin (Carboplatin Injection)
- Adjuvant Radiotherapy (Active Comparator): 1. Histopathological grade G3 and <50% myometrial invasion: Vaginal brachytherapy 5Gy, 3 times;
  2. Histopathological grade G3 and vascular space involvement: Pelvic radiation 45-50 Gy;
  3. ≥50% myometrial invasion: Pelvic radiation 50 Gy + Vaginal brachytherapy 5Gy, 2-4 times.
  Interventions: Radiation: Pelvic Radiation; Radiation: Vaginal Brachytherapy 1; Radiation: Vaginal brachytherapy 2

INTERVENTIONS:
Drug: Paclitaxel — 175 mg/m(2), intravenously (IV)
  Arms: Adjuvant Chemotherapy
Drug: Paraplatin (Carboplatin Injection) — AUC=5, IV
  Arms: Adjuvant Chemotherapy
Radiation: Pelvic Radiation — 45-50 Gy
  Arms: Adjuvant Radiotherapy
Radiation: Vaginal Brachytherapy 1 — 5 Gy, 3 times
  Arms: Adjuvant Radiotherapy
Radiation: Vaginal brachytherapy 2 — 5 Gy, 2-4 times
  Arms: Adjuvant Radiotherapy

SUMMARY:
This randomized trial is studying the efficacy and safety of the chemotherapy compared with radiation therapy alone as adjuvant treatment after operation in Patients with high risk and Stage I endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* FIGO stage: Ⅰ, endometrial carcinoma;
* Female, Chinese women;
* Initial treatment is staging surgery;
* Pathological diagnosis: Endometrial adenocarcinoma;
* Pathologic examination and meet the following one of the indications of adjuvant therapy: ① histopathological grading in poorly differentiated: G3; ② ≥50% myometrial invasion; ③ vascular space involvement;
* No prior treatment;
* Provide written informed consent.

Exclusion Criteria:

* Unable to receive surgery and/or unsuitable for radiotherapy or chemotherapy;
* Family history of ovarian cancer;
* Suffering from other malignancies;
* Concurrently participating in other clinical trials;
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-11; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 3-year DFS

SECONDARY OUTCOMES:
Side effect of adjuvant chemotherapy | 3-month，6-month，1-year and 3-year
  The incidence of infusion reactions (i.e.,skin reactions, cardiovascular reactions, respiratory or throat tightness), and allergic reactions (i.e., life-threatening anaphylaxis)
Complications of radiotherapy | 3-month，6-month，1-year and 3-year
  To observe the subtle effect on quality of life (e.g., diarrhea, bowel symptoms) and vaginal stenosis.
Quality of Life | 3-month，6-month，1-year and 3-year
Overall survival (OS) | 3-year OS

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (3):
- China (3):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang